CLINICAL TRIAL: NCT04120246
Title: A Phase I Dose Escalation Trial of Alpha-Tocopheryloxyacetic Acid (α-TEA) in Patients With Treatment Refractory HER2+ Metastatic Breast Cancer
Brief Title: Alpha-TEA and Trastuzumab for the Treatment of Refractory HER2+ Metastatic Breast Cancer
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Study placed on hold.
Sponsor: Veana Therapeutics (Industry)
Collaborators: University of Washington (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1004302; NCI-2019-06457 (Registry Identifier: NCI / CTRP); 8790 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2019-10-07; First posted 2019-10-09 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; HER2 Positive Breast Carcinoma; Metastatic Breast Carcinoma; Refractory Breast Carcinoma
Keywords: Breast; HER2+; metastatic; refractory; immunotherapy
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — 2,5,7,8-tetramethyl-2R-(4R,8R,12-trimethyltridecyl)chroman-6-yloxy acetic acid; Acetic Acid; Trastuzumab; Antibodies, Monoclonal; PF-05280014; Ogivri; Ontruzant; trastuzumab biosimilar HLX02

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (alpha-TEA, trastuzumab) (Experimental): Patients receive one of 4 doses of alpha-TEA PO on days 1-14 of each cycle. Patients also receive trastuzumab on day 1 of cycle 1 and then every 3 weeks per standard of care. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Alpha-tocopheryloxyacetic Acid; Biological: Trastuzumab

INTERVENTIONS:
Drug: Alpha-tocopheryloxyacetic Acid — Given PO
  Other Names: 12-trimethyltridecyl) chroman-6-yloxy) Acetic Acid; a-TEA; alpha-TEA; 261929-52-6
Biological: Trastuzumab — Given IV
  Other Names: 180288-69-1; 688097; ABP 980; Anti-c-ERB-2; Monoclonal Antibody; Anti-ERB-2; Anti-erbB2 Monoclonal Antibody; Anti-HER2/c-erbB2 Monoclonal Antibody; HER2 Monoclonal Antibody; Herceptin; Herceptin Trastuzumab Biosimilar PF-05280014; Herzuma; MoAb HER2; Monoclonal Antibody HER2; Ogivri; Ontruzant; RO0452317; Trastuzumab Biosimilar ABP 980; Trastuzumab Biosimilar HLX02; Trastuzumab Biosimilar PF-05280014; Trastuzumab Biosimilar SB3; Trastuzumab-DTTB; Trazimera; Kanjinti; Trastuzumab Biosimilar GB221

SUMMARY:
This phase I trial studies the side effects and best dose of alpha-TEA when given together with trastuzumab and to see how well they work for the treatment of HER2+ breast cancer that does not respond to treatment (refractory) and has spread to other places in the body (metastatic). Anti-cancer treatment, such as alpha-TEA, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Alpha-TEA may also alter cancer growth by stimulating the body's immune response against the tumor. Trastuzumab is a form of "targeted therapy" because it works by attaching itself to specific molecules (receptors) on the surface of cancer cells, known as HER2 receptors. When trastuzumab attaches to HER2 receptors, the signals that tell the cells to grow are blocked and the cancer cell may be marked for destruction by the body's immune system. Giving alpha-TEA and trastuzumab may work better for the treatment of HER2+ refractory and metastatic breast cancer compared to usual treatment.

DETAILED DESCRIPTION:
OUTLINE:

This is a dose-escalation study of alpha-TEA.

Patients receive one of 4 doses of alpha-TEA orally (PO) on days 1-14 of each cycle. Patients also receive trastuzumab on day 1 of cycle 1 and then every 3 weeks per standard of care. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months for 4 years.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with HER2/neu overexpressing metastatic breast, not considered curable by conventional therapies

   1. HER2 positivity will be defined per the 2018 ASCO/CAP guidelines (JCO 2018)
   2. Has measurable extra-skeletal disease per RECIST 1.1
2. Patients who have received recommended first therapy with a Taxane, with trastuzumab and/or pertuzumab and second line therapy with Kadcyla (ado-trastuzumab emtansine) or ENHERTU (fam-trastuzumab deruxtecan-nxki) or are unable to tolerate these therapies are eligible to participate.
3. Patients must continue trastuzumab or biosimilars of trastuzumab with or without pertuzumab dosing per standard of care through the entire study period.
4. Prior Lapatinib in the metastatic setting is allowed, but not required.
5. Patients with ER and / or PR positive metastatic breast cancer are eligible and may continue anti-estrogen therapy for the duration of the study.
6. Patients must be at least 14 days post cytotoxic chemotherapy prior to enrollment.
7. Patients on bisphosphonates and/or endocrine therapy are eligible and can continue on this therapy concurrently.
8. Women who are having sex that can lead to pregnancy must have a negative pregnancy test within 28 days prior to enrollment and must avoid becoming pregnant while on α-TEA and for 4 weeks after the last dose of α-TEA and 7 months after Herceptin/biosimilars (see section 7.3). Men must avoid fathering a child while on α-TEA and for 4 weeks after the last dose of α-TEA.
9. Patients must have ECOG Performance Status Score of ≤ 2 (Appendix A).
10. Patients must have recovered from major infections and/or major surgical procedures, and in the opinion of the investigator, not have significant active concurrent medical illnesses precluding study treatment.
11. Laboratory values must be as follows and performed within 28 days prior to first treatment

    1. WBC ≥ 2000/mm3
    2. Hgb ≥ 8 mg/dl
    3. Estimated creatinine clearance (Clcr) by the Cockcroft-Gault (G-C) equation ≥ 60 mL/min
    4. Total bilirubin ≤ 1.5 x upper limit of normal
    5. AST <2.5 X upper limit of laboratory normal
    6. ALT<2.5 X upper limit of laboratory normal
    7. Alkaline phosphatase <2.5 X upper limit of laboratory normal
    8. INR <1.5
    9. PT <16 seconds
    10. PTT < 38 seconds
    11. TSH ≤ 5
    12. Free T4 ≥ .9
12. Ability to swallow capsules.
13. Patients must be at least 18 years of age.
14. Patients must have adequate cardiac function as demonstrated by normal left ventricular ejection fraction (LVEF) ≥ the lower limit of normal for the facility (or ≥50%) on MUGA scan or echocardiogram (ECHO) within 3 months of enrollment.
15. Must be off Vitamin E supplements (multivitamin acceptable) for at least two weeks prior to first dose of study drug

Exclusion Criteria:

* 1. Patients with any of the following cardiac conditions:

  1. Restrictive cardiomyopathy
  2. Unstable angina within 6 months prior to enrollment
  3. New York Heart Association functional class III-IV heart failure
  4. Symptomatic pericardial effusion
  5. Right atrial enlargement on ECHO would not be allowed. 2. History of or active atrial fibrillation or supraventricular tachycardia 3. History of documented cardiac arrhythmia 4. Active cardiac ischemia. Patients with a history of ischemia ameliorated with stent placement or coronary artery bypass grafting and who have no evidence of ischemia by exercise or physiological stress testing are eligible.

     5. Patients with any clinically significant autoimmune disease requiring active treatment.

     6. Patients receiving any concurrent systemic immunosuppressants within 14 days of enrollment. Patients who require brief courses of steroids to manage allergic reaction to intravenous contrast used in radiographic studies are eligible.

     7. Patients receiving strong inhibitors or inducers of CYP3A4/5. (See Appendix B - Patients must be off at least 2 weeks prior to first dose of IP) 8. Patients who are pregnant or breast-feeding. 9. Patients who are simultaneously enrolled in other treatment studies for active treatment.

     10. Active brain metastatic disease. Patients with brain metastases who have been treated with surgery, gamma-knife radiosurgery or radiation and no radiographic progression for at least 4 weeks and off steroids for 14 days are eligible.

     11. No leptomeningeal disease. 12. Any medical or psychiatric condition that in the opinion of the PI would preclude compliance with study procedures.

     13. Malabsorption state such as ulcerative colitis, previous surgical resection of > 20% of intestine or stomach.

     14. Surgery or severe trauma within 4 weeks of study entry (minimally invasive procedures acceptable).

     15. QTc greater than 450 msec at (calculated using Bazett's formula), sick-sinus syndrome or other active cardiac disease.

     16. Patient with abnormal thyroid function or who are euthyroid but on medication for thyroid disorders must be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-04-08 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2030-02-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events of 4 escalating doses of alpha-tocopheryloxyacetic acid (TEA) therapy when combined with trastuzumab | Up to 4 years
  Toxicity grading will be evaluated per Cancer Therapy Evaluation Program (CTEP) Common Terminology Criteria for Adverse Events (CTCAE) 5.0.
Clinical response rate of alpha-TEA when combined with trastuzumab | Up to 4 years
  Clinical response will be performed by computed tomography (CT) scan of the chest, abdomen, and pelvis performed prior to enrollment and then after every 3 cycles per standard of care. Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria and immune related (ir)RECIST criteria will be used to determine response. Both progression free survival (PFS) and overall survival (OS) will be measured.

SECONDARY OUTCOMES:
Change in level of activated effector memory CD4+ and CD8+ T-cells at 4 escalating doses of alpha-TEA and concurrent trastuzumab | At baseline, at cycle 4 Day 1, and then Day 1 of every 4th cycle while on study (each cycle is 28 days), assessed up to 4 years
  The level of memory CD4+ and CD8+ T cells will be evaluated by flow cytometry. Memory CD4+ T cells will be defined as CD3+CD4+CD38+HLA-DR+CCR7-CD45RA- and memory CD8+ T cells will be defined as CD3+CD8+CD38+ HLA-DR+CCR7-CD45RA-.
Change in the number of HER2 specific T cells at each dose level | Baseline up to 4 years
  Will determine if concurrent alpha-TEA and trastuzumab increase the number of HER2 specific T cells at each dose level. Endogenous immunity to HER2 will be evaluated using interferon (IFN)-gamma enzyme-linked immunosorbent spot (ELISPOT) assay. A statistically significant increase of HER2 specific immunity after concurrent alpha-TEA and trastuzumab treatment when compared to baseline will constitute augmentation of HER2 specific immunity.
Modulation of circulating natural killer (NK) cells with concurrent alpha-TEA and trastuzumab therapy | At baseline, at cycle 4 Day 1, and then Day 1 of every 4th cycle while on study (each cycle is 28 days), assessed up to 4 years
  Flow cytometry will be used to assess the number of NK cells as defined by CD3-CD16+CD56+ cells from whole blood. Flow will be used to analyze the function of NK cells, specifically through degranulation markers (CD107a+) and through IFN-gamma production. The level of NK cell CD107+ uptake and IFN-gamma production in response to major histocompatibility complex (MHC) class 1 negative cell will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: William Gwin, MD, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (2):
- United States (2):
  - Providence Cancer Institute - Franz Clinic, Portland, Oregon
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No